CLINICAL TRIAL: NCT03458312
Title: Nurse-led Family and Network Consultations - Addressing Cancer-Related Symptoms and Concerns in Patients With High-grade Glioma and Their Families and Network (CARES)
Brief Title: Nurse-led Family and Network Consultations
Acronym: CARES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: The Novo Nordic Foundation (Other)
Responsible Party: Principal Investigator, Karin Piil, Ph.D. Research and quality manager, Rigshospitalet, Denmark
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CARES
Record Dates: First submitted 2018-01-05; First posted 2018-03-08 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: High-grade Glioma
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Intervention Model Description: To explore the feasibility of a 'Nurse-led Family and Network Consultation' (FNC) that seek to identify and address patients' symptoms/concerns and caregiver burden on one side and identify the resources and opportunities to ease their burdens on the other side.
  To explore the impact of these nurse consultations on the nurses' perception of autonomy, self-esteem, and confidence, representing their professional identity
Masking Description: a sample of patients with HGG (n=30) and their caregivers (n=30) recruited for intervention group (IG) with 'Nurse-led Family and Network Consultations' using pretest and posttest measures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Family and Network support measurements (No Intervention): The perceived 'Family support' and 'Caregiver burden' (FNC) will be measured among 30 families.
  Test time points:
  Post 1. FNC (week 1-2), post FNC 2 (week 8-10) and post FNC 3 (week 28-30) and post the 4. FNC (week 50-52)
- Family and network consultations (Experimental): Intervention: FNC IG will receive four family consultations over 52 weeks relying on the Calgary model and Patient-reported outcome on symptom management and concerns.
  Interventions: Behavioral: Family and Network Consultations

INTERVENTIONS:
Behavioral: Family and Network Consultations — Family and Network Consultation' (FNC) seek to identify and address patients' symptoms/concerns and caregiver burden on one side and identify the resources and opportunities to ease their burdens on the other side.
  Intervention: FNC IG will receive four family consultations over 52 weeks relying on the Calgary model and Patient-reported outcome on symptom management and concerns.
  Arms: Family and network consultations

SUMMARY:
Patients diagnosed with high-grade gliomas (HGG) experience a complex symptom burden including high-levels concerns.

As a consequence to this life-threatening disease, the rely on close contact with a specialized neuro-oncological team as well as support and practical assistance from their families. However, multidimensional burden of caregivers has been reported.

CARES seeks to facilitate and activate the existing resources within the patient and the network using a new model of systematic family care approach.

Specialized neuro-oncological nurses are responsible for an expanded area providing an opportunity for the nursing profession to establish a new model of nursing care. This may not only benefit the patients and their families but also contribute to strengthen the nurses' professional identity and support further development of neuro-oncological specialist team.

DETAILED DESCRIPTION:
Objectives To explore the feasibility and benefits of a 'Nurse-led Family and Network Consultation' (FNC) that seek to identify and address patients' symptoms/concerns and caregiver burden on one side and identify the resources and opportunities to ease their burdens on the other side.

To explore the impact of these nurse consultations on the nurses' perception of autonomy, self-esteem, and confidence, representing their professional identity.

Methods This is a feasibility study in two parts: 1) a sample of patients with HGG (n=30) and their caregivers (n=30) recruited for informing the study about the family function, support and caregiver burden and 2) a sample of patients with HGG (n=30) and their caregivers (n=30) recruited for intervention group (IG) with 'Nurse-led Family and Network Consultations' using pretest and posttest measures.

Part two applies a Mixed Method convergent design with a QUAL + QUAN design.

Nursing BA students at Metropolitan University College will carry out affiliated bachelor projects within CARES.

Theoretical framework Biopsychosocial Model International Classification of Functioning, Disability and Health (ICF) Use of narratives within neuro-oncology Feedback models and goal setting Symptom management theory The integrated Framework of Family System Nursing; Calgary Model Model of levels of personal and professional change

Intervention: FNC IG will receive four family consultations over 52 weeks relying on the Calgary model and Patient-reported outcome on symptom management and concerns.

Measurements

Test time points:

Post 1. FNC (week 1-2), post FNC 2 (week 8-10) and post FNC 3 (week 28-30) and post the 4. FNC (week 50-52).

Part 1, questionnaires for cohort patients (n=30) and caregivers:

The Caregiver Burden Scale (only caregivers) Hospital Anxiety and Depression Scale (HADS),(only caregivers)

The ICE Family Perceived Support Questionnaire (ICE-FPSQ) (caregiver and patient, individually) Psychometric development of the Iceland-Expressive Family Functioning Questionnaire (ICE-EFFQ) (caregiver and patient, individually)

Part 2, questionnaires for IG patients (n=30):

The M.D. Anderson Symptom Inventory-Brain Tumour Module (before FNC) HADS The Functional Assessment of Cancer Therapy-Brain (FACT-Br) ICE-FPSQ ICE-EFFQ

Questionnaires for IG family members (n=30):

The Caregiver Burden Scale HADS ICE-FPSQ ICE-EFFQ

Material from the FNC Written resume of each consultation (n=120)

Interviews:

Semi-structured telephone interviews with IG patients (n=30) and IG family member (n=30) post FNC 2 and post FNC 4 Focus group interview with project nurses post FNC 5 (n= 5 nurses)

Analysis The MDASI-BT, HADS, FACT-Br, the ICE-EFFQ, the ICE-FPSQ and Caregiver burden scale to be analysed separately.

Thematic analyses of interviews, field notes and resume according to Braun and Clarke.

The Mixed Methods analytic approach is interpretive integration, which merges, compares, contradicts and discusses the data sets in order to achieve analytic integration in meta-inference.

Time schedule May 2017 - December 2017: The preparatory phase February 2018 -August 2019: Cohort data collection March 2018- July 2018: Education of the project nurses August 2018 - February 2020: Intervention (1-year intervention with 6 months recruitment)

Clinical and research implications New model of care in expanded nurse-led consultations relying on FNC may be powerful way to facilitate strategies to improve symptom management, emotional well-being and reduce concerns among families.

This study will take at neurosurgical department and oncological department at Copenhagen University Hospital, Rigshospitalet in cooperation with neuro-oncological specialist team.

ELIGIBILITY:
Inclusion Criteria:

-

Patients in the cohort (n=30) and IG (n=30) and their families will be recruited within the first week after surgery. Included are:

* Patients ≥ 18 years of age and newly diagnosed with HGG (WHO classification grade III/IV) after biopsy or operation.
* The patients and their family members and network must be able to speak and understand Danish.
* Provide informed consent

Exclusion Criteria:

* Excluded are • Patients without family or any network. There are no restrictions regarding the family members/network relation to the patient as long as the patient has accepted the person(s) as being a close relative or friend that the patient allows to participate in the FNC. Written informed consent will be obtained before discharge from the hospital or by telephone after discharge.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2018-04-09 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
The experiences from participation in Family and network consultations (FNC) | At week 50 to 52
  Interviews seek the perspectives on the life situation related to the participation of FNC

SECONDARY OUTCOMES:
Change in the perceived Caregiver Burden Scale over time (only caregivers) | At week 1-2, week 8-10, week 28-30 and week 50-52
  Self-reported caregiver burdens. The changes in frequencies will be calculated. No rating scale The scores of the 22 items of the Caregiver Burdenscale will be added together to produce the five sub-scales. The overall mean caregiver burden will be divided into three groups: low burden (1.00-1.99), medium burden (2.00-2.99) and high burden (3.00-4.00).
Change in the severity of depressive symptoms over time measured by the Hospital Anxiety and Depression Scale (HADS) | At week 1-2, week 8-10, week 28-30 and week 50-52
  The self-reported prevalence and severity of depressive symptoms over time. The changes will be presented as separate scores for depressive symptoms.
  higher scores indicating greater likelihood of depression or anxiety.
Change in the severity of anxiety over time measured by the Hospital Anxiety and Depression Scale (HADS) | At week 1-2, week 8-10, week 28-30 and week 50-52
  The self-reported prevalence and severity of anxiety over time. The changes will be presented as separate scores for depressive symptoms.
  higher scores indicating greater likelihood of depression or anxiety.
Changes in the perception of received support from nurses will be measured by the ICE Family Perceived Support Questionnaire (ICE-FPSQ) (caregiver and patient, individually) | At week 1-2, week 8-10, week 28-30 and week 50-52
  Changes in Support from nurses. No rating scale.
The perceived changes of the functioning within a Family will be measured by the Psychometric development of the Iceland-Expressive Family Functioning Questionnaire (ICE-EFFQ) (caregiver and patient, individually) | At week 1-2, week 8-10, week 28-30 and week 50-52
  Changes in Family Functioning. No rating scale.
The prevalence of symptoms over time will be measured by the M.D. Anderson Symptom Inventory-Brain Tumour Module | At week 1-2, week 8-10, week 28-30 and week 50-52
  Changes in Symptoms will be reported. Each symptom is rated on a 0-10 scale (0 = ''not present'' and 10 = ''as bad as you can imagine'') over the past 24 hours. Six interference items assessing symptom-related interference in general activity, mood, work (including work around the house), relations with other people, walking, and enjoyment of life also are included in the MDASI. Each interference item is rated on a 0e10 scale (0 = ''did not interfere'' and 10 = ''interfered completely'') over the past 24 hours.
The quality of life will be measured by The Functional Assessment of Cancer Therapy-Brain (FACT-Br) | At week 1-2, week 8-10, week 28-30 and week 50-52
  The self-reported quality of life related to brain cancer is measured by FACT-G. It comprises 4 sub-scales: physical well-being (PWB), social/family well-being (SWB), emotional well-being (EWB) and functional wellbeing (FWB), on a 5-point Likert scale ranging from 0 (not at all) to 4 (very much). Moreover, the brain cancer sub-scale (BrCS) reflects issues specific for brain cancer. The highest possible score is 28 for the PWB, SWB and FWB subscales, 24 for the EWB subscale and 184 for the BrCS. FACT-Br total score is the sum of the 4 sub-scales (of the core instrument). The FACT-G total score provides a summary of the overall HRQOL across the group of patients [range 0-108] and the FACT-Br Trial Outcome Index [range 0-132] is a summary index of physical/functional outcomes. The higher the score, the better HRQOL.

OTHER OUTCOMES:
Change in the perception of the nurses professional identity | At week 28-30 and week 50-52
  Change in Professional identity

CONTACTS AND LOCATIONS:
Locations (1):
- University hospital of Copenhagen, Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Piil K, Laegaard Skovhus S, Tolver A, Jarden M. Neuro-Oncological Symptoms: A Longitudinal Quantitative Study of Family Function, Perceived Support, and Caregiver Burden. J Fam Nurs. 2022 Feb;28(1):43-56. doi: 10.1177/10748407211029986. Epub 2021 Jul 21. PMID 34286624